CLINICAL TRIAL: NCT05289141
Title: Interest in the Use of Nasal High-Flow Oxygen Therapy (OptiFlow™) in Secondary Transport of COVID-19 Positive Patients
Acronym: SAMU83
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-CHITS-002
Record Dates: First submitted 2022-03-18; First posted 2022-03-21 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: Coronavirus disease 2019 (COVID-19); Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); Nasal High-Flow Oxygen Therapy; Secondary transport by emergency medical service; Non-invasive ventilation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated by high flow nasal oxygen therapy (Optiflow™)
  Interventions: Device: Use of high flow nasal oxygen therapy
- Patients treated by other non-invasive ventilation or high concentration oxygen masks
  Interventions: Device: Use of other non-invasive ventilation or high concentration oxygen masks

INTERVENTIONS:
Device: Use of high flow nasal oxygen therapy — Use of high flow nasal oxygen therapy during secondary transport by emergency medical service 83 (SAMU 83).
  Groups: Patients treated by high flow nasal oxygen therapy (Optiflow™)
Device: Use of other non-invasive ventilation or high concentration oxygen masks — Use of other non-invasive ventilation or high concentration oxygen masks during secondary transport by emergency medical service 83 (SAMU 83).
  Groups: Patients treated by other non-invasive ventilation or high concentration oxygen masks

SUMMARY:
Since the beginning of COVID-19 pandemic situation, several modes of ventilation have been tried to correct the hypoxaemia induced by SARS-CoV-2 virus. A few recent studies have concluded that high-flow nasal oxygen therapy (OptiFlow™) is beneficial in COVID-19. All mainly conclude that the use of OptiFlow™ avoid intubations and decrease hospitalization duration in critical care services.

At the emergency medical service 83 (SAMU 83), it has been decided to extend this ventilation mode during patient secondary transfers (transfer from an intensive care unit/other hospital unit/emergency department to another hospital's intensive care unit).

The emergency medical service 83 has equipped its intensive-care ambulances with OptiFlow™ in order not to interrupt this ventilation mode during transport.

The hypothesis is that patients with a severe respiratory form of COVID-19 transported from one health facility to another by the emergency medical service 83 on high-flow nasal oxygen therapy has a reduced risk of intubation compared to the other modes of non-invasive ventilation (NIV) and High Concentration oxygen Masks (HCM).

DETAILED DESCRIPTION:
Retrospective observational study in France including COVID-19 infected patients taken care of by the emergency medical service 83 (SAMU 83) for a secondary transport between1st March 2020 and 31th December 2021.

ELIGIBILITY:
Inclusion Criteria:

* COVID-positive patient diagnosed either by positive Polymerase Chain Reaction (PCR) or radiological interpretation of chest CT
* Patient in respiratory distress treated during transport by high flow nasal oxygen or HCM (with a minimum flow of 15 L/min) or other NIV modes
* Patient taken care of by the emergency medical service 83 (SAMU 83) for secondary transport (transfer from an intensive care unit/other hospital unit/emergency department to another hospital's intensive care unit) between1st March 2020 and 31th December 2021

Exclusion Criteria:

* Pre-transport intubation
* Patient opposition to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients more than 18 year old taken care of by the emergency medical service 83 (SAMU 83) for secondary transport (transfer from an intensive care unit/other hospital unit/emergency department to another hospital's intensive care unit) between1st March 2020 and 31th December 2021 and without pre-transport intubation
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Intubation rate | 24 hours
  Rate of intubation during the first 24 hours after arrival in the destination Intensive Care Unit (ICU)

SECONDARY OUTCOMES:
Mortality rate | 28 days
  Rate of patients alive at Day 28.
ICU length of stay | At the moment of Intensive care unit discharge, up to 1 month
  Number of days spent in intensive care unit of destination

CONTACTS AND LOCATIONS:
Overall Officials: BOUTIN Célia, MD, Study Director — Centre Hospitalier Intercommunal Toulon - La Seyne sur Mer
Locations (1):
- Centre Hopitalier Intercommunal Toulon - La Seyne sur Mer, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No